CLINICAL TRIAL: NCT02307552
Title: Transurethral Ultrasonic Imaging For Detection and Classification of Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The probe could not be anchored in place and would rotate about its axis, thus comparison was difficult.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Thomas E. Ahlering, Vice Chairman and Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-9305
Record Dates: First submitted 2014-08-28; First posted 2014-12-04 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Imaging; ultrasound; prostate; cancer; diagnostic tool; catheter; urethra; digital rectal exam
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All patients in the study will receive a scan of their prostate with the novel UreScan machine. All scans will be evaluated in their accuracy of detecting cancer loci within the prostate as compared to histopathological reviews of the prostate post robotic prostatectomy.
  Interventions: Device: UreScan

INTERVENTIONS:
Device: UreScan — The TUUS Foley/catheter will be inserted into the urethra via the ultrasound visualization onto the apex prostate, and the ultrasound extended through the urethra until the bladder neck and stopped. This is recorded twice automatically, and this should take 5-10 minutes for completion, and the prostate ultrasound data stored in memory. The ultrasound/subject interaction is now complete, and the study should add 30-60 minutes to the preoperative visit. No local or general anesthesia is used. The subject will be given 500 mg of Ciprofloxacin as a preventative measure against a urinary tract infection.

SUMMARY:
This study is being performed to verify the ability to use minimally invasive transurethral ultrasonic imaging technology for the purpose of identifying prostate cancer. Transurethral ultrasonic prostate imaging, may in the future, be used for detection and monitoring these disease processes to minimize the need for obtaining surgical biopsy specimens. The hypothesis is that tissue-density variations, as revealed in diagnostic ultrasonic imaging, results in unique image signatures for identification of prostate cancer. This imaging procedure provides a multifaceted view of the entire in-situ gland.

The current use of Prostate Specific Antigen (PSA) for determining the likelihood of presence of cancer in the prostate gland requires interpretation and has a good but limited to predict prostate cancer on biopsy, with significant false prediction rates. More importantly as a blood test, the PSA test lacks the ability to pinpoint the location of the cancer within the prostate gland. Preliminary study findings have suggested that "Transurethral Ultrasonic Scanning" (TUUS) presents the desired improved diagnostic sensitivity for detection of cancer within the imaged prostate gland, and has the intrinsic capability to provide high resolution images of the transverse and future three-dimensional views of the entire gland better than currently used Transurethral Ultrasound (TRUS). Two important goals of the practicality of this minimally invasive technology will be assessed by this study. 1. The ability of TUUS to directly detect prostate cancer locations in the prostate. 2. The use of TUUS to successfully guide the prostate needle biopsy to cancer loci with a high rate accuracy.

DETAILED DESCRIPTION:
The Purpose of the Research The primary objective of this Institutional Review Board-controlled study is to determine if the presently manually-read results of TUUS data obtained with the novel UreScan device can be correlated with pathologist findings in a harvested prostate gland from an individual with diagnosed prostate disease. If successful, a future Institutional Review Board study will explore the use of computer software to examine the 256 transverse image slices of a large number of prostate cancer patients to establish the clinical applicability of TUUS for screening and assessment of individuals with elevated levels of PSA and/or positive digital rectal examinations (DRE), potentially reducing the number of future biopsy examinations with false-positive findings.

Background Information The current use of Prostate Specific Antigen for determining the likelihood of presence of cancer in the prostate gland has been shown to be seriously flawed. Multiple studies reviewing the findings of referred biopsies, based on elevated PSA levels, resulted in as many as 70% false positive findings for cancer. Improved rapid, minimally-invasive, low-cost methodology and technology should be developed to provide diagnostic cancer findings that have higher sensitivity and specificity is the objective goal of the present research. Preliminary study findings have suggested that "Transurethral Ultrasonic Scanning" (TUUS) presents the desired improved diagnostic sensitivity for detection of cancer within the imaged prostate gland and has the intrinsic capability to provide high resolution images of the transverse and future three-dimensional views of the entire gland. Two important goals of this minimally invasive technology will be assessed by this study. 1. The ability of TUUS to directly detect prostate cancer in situ in the prostate. 2. The use of TUUS to successfully guide the prostate needle biopsy to cancer loci with a high rate accuracy.

In a 2003 study by Holmes et al, the TUUS device was tested on 2 patients who had seeds implanted for prostate cancer. TUUS revealed more seeds (82%, 84%) than standard TRUS (63%, 65%) in the 2 patients. These simple cases demonstrated the feasibility of providing transverse images of the entire prostate gland. Holmes postulated that this procedure would have to be automated to achieve any clinical utility value and the project essentially was abandoned by Mayo.

The TUUS/"UreScan" system is a marriage of an off label usage of the FDA approved vascular probe, placed inside a standard foley catheter which is inserted into the penis onto the prostate to the neck of the bladder. The ultrasound probe travels the length of the prostate (~4-8cm) within the sheath of the catheter and images the entire prostate with ultrasound. The travel of the ultrasound probe is controlled by a small motor which is driven from outside the catheter and patient as well. This motor driven probe offers the possibility of accurate and reproducible ultrasounds of the prostate, as the patient's prostate apex is used the anchor point for study.

Refinements to the TUUS system include:

1. A Foley type introducer should be used for placing the intravascular ultrasound transducer in the prostatic urethral region to be imaged
2. Use of a fixed-position, ultrasonic coupling gel-coated Introducer to eliminate the possibility of urethral abrasion or trauma as might otherwise occur without the Introducer when moving the transducer within the prostatic imaging region.
3. Insertion into the Introducer of the wire-rotationally-driven ultrasonic transducer as coated with sterile water ultrasonic coupling between the transducer and introducer
4. The examiner would then initiate the automated scanning procedure with analog/digital video data for each of 256 transverse axial image slices of the prostate gland. The scanning of the gland can be stopped or started at the election of the examiner
5. A video-media record of the images derived from the procedure is available to an experienced reader for interpretation.

The initial UreScan hydrophone verified specifications included: 1. 256 transverse, automatically axially advanced, image slices. 2. Approximately 267 megabits of video data. 3. Diagnostic ultrasound scanning of 100 revolutions per minute at 9.0 M Megahertz. 4. Radial penetration of 6 cm. The scanner features:

1. The amplitude of reflected ultrasonic echoes from biological tissue, as displayed by a density-based oscillogram is directly proportional to the density of the tissue being insonated in an adjusted flat far-gain ultrasonic system.
2. Longitudinal time-related, ultrasonic densitometry and image-registered comparisons of sonograms have demonstrated progression and/or regression of disease consistent with efficacy of treatment procedures. This facilitates future "wait and watch surveillance" of known or suspected lesions while potentially minimizing and/or eliminating unnecessary surgical biopsy tissues procedures
3. The reflected echo waveform and sonogram has been shown to be unique for each type of disease entity. In prostate disease, there is a unique difference between the image-markers for prostate cancer and normal tissue.

The present study protocol is to determine if image-markers for cancer and other unique prostate pathology can be specifically identified. Further clinical studies will be required to determine sensitivity, specificity, accuracy and (+/-) predictor values of this procedure. Additional studies will be required to determine if the amplitude of the image-markers could be used for determining the approximate stage of the image detected disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing a standard of care radical prostatectomy for prostate cancer.
* Aged > 40 years old.
* Men who have a serious prostate obstruction, are excluded due to the difficulty of catheter insertion.

Exclusion Criteria:

* Women are excluded as they do not have a prostate gland.
* Minors are excluded as prostate cancer is generally found only in men aged > 40 years old

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Ahlering, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Health, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holmes DR 3rd, Davis BJ, Bruce CJ, Robb RA. 3D visualization, analysis, and treatment of the prostate using trans-urethral ultrasound. Comput Med Imaging Graph. 2003 Sep-Oct;27(5):339-49. doi: 10.1016/s0895-6111(02)00102-7. PMID 12821027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1
Arm/Group | All Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure Novel Transurethral Ultrasound Signatures to Detect Prostate Cancer
Description: The primary objective of this Institutional Review Board -controlled study is to determine if Trans urethral ultrasound can be used to identify prostate cancer, thus avoiding prostate needle biopsies for diagnosis
Time Frame: one year
Population: Data were not collected because the study was discontinued due to lack of feasibility and negative results.
Arm/Group | All Patients
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No